CLINICAL TRIAL: NCT05518136
Title: APP Rehabilitation Management and Evaluations of Cardiopulmonary Function and Motor Development in Infants With Congenital Heart Disease: a Pilot Study
Brief Title: Evaluations of Cardiopulmonary Function and Motor Development of Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gejingwa Zhao (Other)
Responsible Party: Sponsor-Investigator, Gejingwa Zhao, Doctor, Doctor of Cardiac Surgery Department, Principal Investigator, Beijing Children's Hospital
Organization: Beijing Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Beijing Children's Hospital
Record Dates: First submitted 2022-08-18; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Congenital Heart Disease in Children; Infant Development; Infant Conditions; Motor Neuropathy; Motor Delay; Cardiopulmonary
Keywords: infant; rehab management APP; home-based exercise; cardiopulmonary endurance; motor developmental level
MeSH Terms: conditions — Neuritis; Psychomotor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery group (Experimental): Recovery group was given home-based rehab exercise periodically supervised by cellphone APP. Left ventricular ejection fractions (LVEF), the rate of increase in heart rate (rHRI), and the rate of recovery heart rate (rHRR) were measured for representing cardiopulmonary capacity. The Alberta test and Neuro-intelligence Scale were used to evaluate their motor developmental outcomes.
  Interventions: Behavioral: exercise-guidance on rehab APP
- Control group (No Intervention): General post-operative care for control group. Left ventricular ejection fractions (LVEF), the rate of increase in heart rate (rHRI), and the rate of recovery heart rate (rHRR) were measured for representing cardiopulmonary capacity. The Alberta test and Neuro-intelligence Scale were used to evaluate their motor developmental outcomes.

INTERVENTIONS:
Behavioral: exercise-guidance on rehab APP — Training motions included sitting balance, hand support, crawling and squatting training12-14 were scheduled for 1 to 3 months postoperatively, moreover, climbing over obstacles was for 3 to 6 months.
  Arms: Recovery group

SUMMARY:
In this single-center, randomized controlled trial, patients (4-8 months) with CHD were randomly assigned to either a recovery group (home-based rehab exercise periodically) supervised by cellphone APP or to a control group. Left ventricular ejection fractions (LVEF), the rate of increase in heart rate (rHRI), and the rate of recovery heart rate (rHRR) were measured for representing cardiopulmonary capacity. The Alberta test and Neuro-intelligence Scale were used to evaluate their motor developmental outcomes. This study verified the feasibility of this rehab method and indicated that 6-month home-based exercise training can improve cardiopulmonary endurance and motor developmental level in infant CHD patients.

ELIGIBILITY:
Inclusion Criteria:

* CHD infants (aged 4-8 months) with atrial septum defect (ASD) or ventricular septum defect (VSD)

Exclusion Criteria:

* chromosomal abnormalities; family history of mental retardation; small for gestational age and prematurity; history of perinatal asphyxia and hyperbilirubinemia; history of central nervous system disease or imaging suggestive of brain dysplasia

Ages: 4 Months to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Baseline LVEF | pre-operative for baseline assessment
  Left ventricular ejection fraction before surgery
Baseline rHRI | pre-operative for baseline assessment
  The rate of increase in heart rate before surgery
Baseline rHRR | pre-operative for baseline assessment
  The rate of recovery heart rate before surgery
Baseline Alberta score | pre-operative for baseline assessment
  Alberta motor test results before surgery
Baseline Neuro-intelligence Scale | pre-operative for baseline assessment
  Developmental Quotient (DQ) before surgery
LVEF one month after the surgery | one month after surgery
  Left ventricular ejection fraction one month after the surgery
rHRI one month after the surgery rHRI one month after the surgery | one month after surgery
  The rate of increase in heart rate one month after the surgery
rHRR one month after the surgery | one month after surgery
  The rate of recovery heart rate one month after the surgery
Alberta score one month after the surgery | one month after surgery
  Alberta motor test results one month after the surgery
Neuro-intelligence Scale one month after the surgery | one month after surgery
  Developmental Quotient (DQ) one month after the surgery
LVEF three months after the surgery | three months after surgery
  Left ventricular ejection fraction three months after the surgery
rHRI three months after the surgery | three months after surgery
  The rate of increase in heart rate three months after the surgery
rHRR three months after the surgery | three months after surgery
  The rate of recovery heart rate three months after the surgery
Alberta score three months after the surgery | three months after surgery
  Alberta motor test results three months after the surgery
Neuro-intelligence Scale three months after the surgery | three months after surgery
  Developmental Quotient (DQ) three months after the surgery
LVEF six months after the surgery | six months after surgery
  Left ventricular ejection fraction six months after the surgery
rHRI six months after the surgery | six months after surgery
  The rate of increase in heart rate six months after the surgery
rHRR six months after the surgery | six months after surgery
  The rate of recovery heart rate six months after the surgery
Alberta score six months after the surgery | six months after surgery
  Alberta motor test results six months after the surgery
Neuro-intelligence Scale six months after the surgery | six months after surgery
  Developmental Quotient (DQ) six months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gejingwa Zhao, Principal Investigator — Beijing Children's Hospital
Locations (1):
- Beijing Children's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gurvitz M, Valente AM, Broberg C, Cook S, Stout K, Kay J, Ting J, Kuehl K, Earing M, Webb G, Houser L, Opotowsky A, Harmon A, Graham D, Khairy P, Gianola A, Verstappen A, Landzberg M; Alliance for Adult Research in Congenital Cardiology (AARCC) and Adult Congenital Heart Association. Prevalence and predictors of gaps in care among adult congenital heart disease patients: HEART-ACHD (The Health, Education, and Access Research Trial). J Am Coll Cardiol. 2013 May 28;61(21):2180-4. doi: 10.1016/j.jacc.2013.02.048. Epub 2013 Mar 28. PMID 23542112

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT05518136/Prot_SAP_000.pdf